CLINICAL TRIAL: NCT02652780
Title: Randomized, Double-Masked, Sham-Controlled Clinical Trial to Evaluate the Efficacy of a Single Intravitreal Injection of GS010 in Subjects Affected for More Than 6 Months and To 12 Months by LHON Due to the G11778A Mutation in the ND4 Gene
Brief Title: Efficacy Study of GS010 for Treatment of Vision Loss From 7 Months to 1 Year From Onset in LHON Due to the ND4 Mutation (REVERSE)
Acronym: REVERSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-LHON-CLIN-03B; 2015-001266-26 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Optic, Atrophy, Hereditary, Leber
Keywords: Leber Hereditary Optic Neuropathy; Leber Hereditary Optic Atrophy; Heredity Optic Atrophy; Eye Diseases; Hereditary Eye Diseases; Inborn Genetic Disease; Genetic Therapy; Intravitreal Injections; Mitochondrial Disease; AAV2 Vectors; Nervous System Diseases; Neurodegenerative Disease; Heredodegenerative Disorders of the Nervous System
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Eye Diseases; Eye Diseases, Hereditary; Genetic Diseases, Inborn; Mitochondrial Diseases; Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GS010-treated Eyes (Experimental): Each participant will have one eye randomly selected to receive a single injection of GS010 and the other eye will receive a sham injection. GS010-treated Eyes: GS010 is a recombinant adeno-associated viral vector serotype 2 (rAAV2/2) containing the wild-type ND4 gene (rAAV2/2-ND4). Participants will receive a single dose of GS010 in one of their randomly selected eyes, via intravitreal injection containing 9E10 viral genomes in 90μL balanced salt solution (BSS) plus 0.001% Pluronic F68®.
  Interventions: Biological: GS010
- Sham-treated Eyes (Sham Comparator): Each participant will have one eye randomly selected to receive GS010 and the other eye will receive a sham injection. Eyes receiving sham injection will undergo the same preparatory procedures as eyes receiving GS010 injection, including pupillary dilation, topical anti-infection and topical anesthetic procedures. Sham Intravitreal injection will be performed by applying pressure to the eye at the location of a typical intravitreal injection procedure using the blunt end of a syringe without a needle.
  Interventions: Device: Sham Intravitreal Injection

INTERVENTIONS:
Biological: GS010 — Both eyes of each participant will receive standard antiseptic preparation, administration of topical local ocular anesthetic agents and will undergo pupillary dilation. Administration of an intra-ocular pressure lowering agent will precede treatment for every participant.
  GS010-treated Eyes: GS010 is a recombinant adeno-associated viral vector serotype 2 (rAAV2/2) containing the wild-type ND4 gene (rAAV2/2-ND4). Participants will receive a single dose of GS010 in one of their randomly selected eyes, via intravitreal injection containing 9E10 viral genomes in 90μL balanced salt solution (BSS) plus 0.001% Pluronic F68®.
  Other Names: Lenadogene Nolparvovec; rAAV2/2-ND4
  Arms: GS010-treated Eyes
Device: Sham Intravitreal Injection — Both eyes of each participant will receive standard antiseptic preparation, administration of topical local ocular anesthetic agents and will undergo pupillary dilation. Administration of an intra-ocular pressure lowering agent will precede treatment for every participant.
  Sham-treated Eyes: One eye of each participant will undergo sham injection. Sham Intravitreal injection will be performed by applying pressure to the eye at the location of a typical intravitreal injection procedure using the blunt end of a syringe without a needle.
  Arms: Sham-treated Eyes

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of GS010, a gene therapy, in improving the visual outcome in participants with Leber Hereditary Optic Neuropathy (LHON) due to the G11778A ND4 mitochondrial mutation when vision loss is present for more than six months and up to one year.

ELIGIBILITY:
Inclusion Criteria:

Selection Criteria:

Participants must meet all the following criteria at the Screening Visit (Visit 1) in order to be included into the study.

1. Age 15 years or older.
2. Onset of vision loss based on medically documented history or participants testimony, in both eyes for 181 and ≤365 days in duration.
3. Each eye of the participant maintaining visual ability to allow at least for counting of the examiner's fingers at any distance.
4. Female participants (if of childbearing potential) must agree to use effective methods of birth control up to 6 months after IVT injection and male participants must agree to use condoms for up to 6 months after IVT injection.
5. Ability to obtain adequate pupillary dilation to permit thorough ocular examination and testing.
6. Signed written informed consent.

Inclusion Criteria:

Participants included in the study must satisfy all the following criteria at the Inclusion Visit (Visit 2).

1. Documented results of genotyping showing the presence of the G11778A mutation in the ND4 gene and the absence of the other primary LHON-associated mutations (ND1 or ND6) in the participant's mitochondrial DNA.
2. Review of all selection criteria to ensure continued compliance.
3. Have a negative test for infection with human immunodeficiency virus (HIV).
4. Have a negative pregnancy test for women of childbearing potential (a woman who is two years post-menopausal or surgically sterile is not considered to be of childbearing potential).

Exclusion Criteria:

Non-Selection Criteria:

Participants who meet at least one of the following criteria at the Screening Visit (Visit 1) will not be included into the study.

1. Any known allergy or hypersensitivity to GS010 or its constituents.
2. Contraindication to IVT injection.
3. IVT drug delivery to either eye within 30 days prior to the Screening Visit (Visit 1).
4. Previous vitrectomy in either eye.
5. Narrow angle in either eye contra-indicating pupillary dilation.
6. Presence of disorders of the ocular media, such as the cornea and lens, which may interfere with visual acuity and other ocular assessments during the study period.
7. Vision disorders, other than LHON, involving visual disability or with the potential to cause further vision loss during the trial period.
8. Causes of optic neuropathy other than LHON and glaucoma.
9. Participants with known mutations of other genes involved in pathological retinal or optic nerve conditions.
10. Presence of ocular or systemic disease, other than LHON, whose pathology or associated treatments might affect the retina or the optic nerve.
11. History of amblyopia associated with a Snellen visual acuity equivalent of worse than 20/80 (equivalent to 6/24 at 6 meters, decimal acuity 0.25, LogMAR +0.6) in the affected eye.
12. Presence of ocular conditions, which in the opinion of the Investigator will prevent good quality SD-OCT imaging from being obtained.
13. Presence, in either eye, of uncontrolled glaucoma, defined as an IOP greater than 25 mmHg, despite maximal medical therapy with intraocular pressure (IOP)-lowering agents.
14. Active ocular inflammation or history of idiopathic or autoimmune-associated uveitis.
15. Participants participating in another clinical trial and receiving an IMP within 90 days prior to the Screening Visit (Visit 1).
16. Previous treatment with an ocular gene therapy product.
17. Participants who have undergone ocular surgery of clinical relevance (per Investigator opinion) within 90 days preceding the Screening Visit (Visit 1).
18. Female participants who are or who intend to breast feed during the trial period.

Exclusion Criteria:

Participants who meet at least one of the following criteria at the Inclusion Visit (Visit 2) will not be included in the study.

1. Any non-selection criteria which may have appeared after the screening visit.
2. Participants taking idebenone who have not completely discontinued the idebenone at least 7 days prior to Visit 2. If the participant has not discontinued idebenone at least 7 days prior to Visit 2, the visit may be delayed until the 7-day period is complete.
3. Presence, at the time of study inclusion, of infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye.
4. Presence of systemic illness, including alcohol and drug abuse (except nicotine), or medically significant abnormal laboratory values that are deemed by the Investigator to preclude the participant's safe participation in the study.
5. Presence of illness or disease that, in the opinion of the Investigator, include symptoms and/or the associated treatments that can alter visual function, for instance cancers or pathology of the central nervous system.
6. Any medical or psychological condition that, in the opinion of the Investigator, may compromise the safe participation of the participant in the study or would preclude compliance with the study protocol or ability of the participant to successfully complete the study.
7. Participants unable or unwilling to comply with the protocol requirements.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yu Wai Man, MDPhDFRCOpht, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (7):
- United States (3):
  - Doheny Eye Center, University of California, Los Angeles, Los Angeles, California
  - Department of Ophthalmology, Emory University School of Medicine, Atlanta, Georgia
  - Neuro Ophthalmologic Associates, Wills Eye Hospital, Thomas Jefferson University, Philadelphia, Pennsylvania
- Centre National Hospitalier d'Ophtalmologie des Quinze-Vingt, Paris, France
- Department of Neurology, University of Munich, Friedrich-Baur-Institute, Munich, Germany
- IRCCS Istituto delle Scienze Neurologiche di Bologna, UOC Clinica Neurologica, Ospedale Bellaria, Bologna, Italy
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carelli V, Newman NJ, Yu-Wai-Man P, Biousse V, Moster ML, Subramanian PS, Vignal-Clermont C, Wang AG, Donahue SP, Leroy BP, Sergott RC, Klopstock T, Sadun AA, Rebolleda Fernandez G, Chwalisz BK, Banik R, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA; the LHON Study Group. Indirect Comparison of Lenadogene Nolparvovec Gene Therapy Versus Natural History in Patients with Leber Hereditary Optic Neuropathy Carrying the m.11778G>A MT-ND4 Mutation. Ophthalmol Ther. 2023 Feb;12(1):401-429. doi: 10.1007/s40123-022-00611-x. Epub 2022 Nov 30. PMID 36449262
- [Derived] Newman NJ, Yu-Wai-Man P, Carelli V, Biousse V, Moster ML, Vignal-Clermont C, Sergott RC, Klopstock T, Sadun AA, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA. Intravitreal Gene Therapy vs. Natural History in Patients With Leber Hereditary Optic Neuropathy Carrying the m.11778G>A ND4 Mutation: Systematic Review and Indirect Comparison. Front Neurol. 2021 May 24;12:662838. doi: 10.3389/fneur.2021.662838. eCollection 2021. PMID 34108929
- See also: National Library of Medicine's Genetics Home Reference for Leber Hereditary Optic Neuropathy — http://ghr.nlm.nih.gov/condition/leber-hereditary-optic-neuropathy
- See also: National Library of Medicine's Genes and Gene Therapy — https://www.nlm.nih.gov/medlineplus/genesandgenetherapy.html

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants who were enrolled and received both study treatments, GS010 and Sham. All participants in the study received both GS010 and the sham procedure simultaneously. Participants were randomly assigned to receive GS010 in either the right or left eye. The same participants also received the sham procedure in the eye not assigned to GS010, at the same study visit.
  GS010: Either the right or left eye received one single dose of GS010 (9E10 vg/eye) via an intravitreal (IVT) injection. The volume of the injected formula was 90 µL. The injection was performed in the vitreous humor under local anesthesia.
  Sham procedure: Either the right or left eye (the eye not randomly assigned to GS010) received the sham procedure. One single sham IVT injection was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
Period: Overall Study
Arm/Group | All Participants
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 32
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
  United Kingdom | 2
  France | 5
  Germany | 6
  Italy | 4
Weight [Mean (Standard Deviation); unit: kilograms] | 80.1 (21.0)
Height [Mean (Standard Deviation); unit: centimetres] | 174.4 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ETDRS Visual Acuity (Quantitative Score) at Week 48
Description: Visual acuity was derived from the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The visual acuity logarithm of the minimal angle of resolution (LogMAR) score was derived from the number of letters participants could read on the ETDRS chart.
  1 ETDRS line = 5 letters
  1 ETDRS line = 0.1 LogMAR
  A lower LogMAR score denotes better visual acuity and a negative change from baseline indicates an improvement in visual acuity.
  Change = (Week 48 score - Baseline score).
Time Frame: Baseline and Week 48
Population: All participants and all eyes that received study treatments, with data at both Baseline and the applicable post-dose visit (Week 48). All participants received both GS010 and Sham simultaneously.
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Units Other Than Participants: Eyes
Groups:
- GS010-treated Eyes: All eyes that received the study treatment, GS010. Each participant was randomly assigned GS010 in either the right or left eye. The eye assigned to GS010 received one single dose of GS010 (9E10 vg/eye) via an intravitreal (IVT) injection. The volume of the injected formula was 90 μL. The injection was performed in the vitreous humor under local anesthesia.
  The same participants also received the sham procedure in the right or left eye, which was not assigned to receive GS010, at the same study visit.
- Sham-treated Eyes: All eyes that received the Sham. Each participant was randomly assigned GS010 in either the right or left eye, the eye not assigned GS010 received the sham procedure. The eye assigned to the Sham received one single sham intravitreal (IVT) injection, which was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
  The same participants also received GS010 in the right or left eye, which did not receive the Sham, at the same study visit.
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
LogMAR | -0.219 (0.055) | -0.211 (0.055)
Statistical Analysis 1: Comparison: GS010-treated Eyes vs Sham-treated Eyes; A mixed model of analysis of covariance (ANCOVA) was used with change from baseline at Week 48 as the response, and participants, eyes of the participant as random factor, treatment and baseline LogMAR value as covariates in the model. P-value is used to assess the significance of the difference between All-GS010 and All-Sham with respect to change of LogMAR from baseline; Test type: Superiority; p = 0.8783, ANCOVA; Mean Difference (Net) = -0.008, 95% CI 2-sided [-0.119 to 0.102]

2. Secondary Outcome: Change From Baseline in ETDRS Visual Acuity (Quantitative Score) at Week 96
Description: Visual acuity was derived from the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The visual acuity logarithm of the minimal angle of resolution (LogMAR) score was derived from the number of letters participants could read on the ETDRS chart.
  1 ETDRS line = 5 letters
  1 ETDRS line = 0.1 LogMAR
  A lower LogMAR score denotes better visual acuity and a negative change from baseline indicates an improvement in visual acuity.
  Change = (Week 96 score - Baseline score).
Time Frame: Baseline and Week 96
Population: All participants and all eyes that received study treatments, with data at both Baseline and the applicable post-dose visit (Week 96). All participants received both GS010 and Sham simultaneously.
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Groups:
- Sham-treated Eyes: All eyes that received the Sham. Each participant was randomly assigned GS010 in either the right or left eye, the eye not assigned GS010 received the sham procedure. The eye assigned to the Sham received one single sham intravitreal (IVT) injection, which was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
  The same participants also received GS010 in the right or left eye, which did not receive the sham procedure, at the same study visit.
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 37
LogMAR | -0.308 (0.068) | -0.259 (0.068)

3. Secondary Outcome: Number of Eye Responders to Treatment at Week 48 and Week 96
Description: An eye was determined as a responder to treatment based on 2 different definitions.
  Definition 1: An eye responder was defined by an improvement of the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score of at least 15 letters compared to Baseline, or a final visual acuity greater than a Snellen acuity equivalent of 20/200 (a score of at least 1 letter).
  Definition 2: An eye responder was defined by an improvement of the ETDRS score of at least 20 letters compared to Baseline.
Time Frame: Baseline; Week 48 and Week 96
Population: All participants and all eyes that received study treatments, with data at both Baseline and the applicable post-dose visit (Week 48 or Week 96). All participants received both GS010 and Sham simultaneously.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes
  Definition 1: Week 48 | 7 | 5
  Definition 1: Week 96 | 12 | 6
  Definition 2: Week 48 | 10 | 13
  Definition 2: Week 96 | 17 | 19

4. Secondary Outcome: Number of Subject Responders to Treatment at Week 48 and Week 96
Description: A subject responder was defined as a participant whose Early Treatment Diabetic Retinopathy Study (ETDRS) score of the treated eye (that received GS010), was at least 15 letters better than the sham eye, or whose treated eye had a logarithm of the minimal angle of resolution (logMAR) acuity score of at least 0.3 logMAR better than the sham eye.
Time Frame: Week 48 and Week 96
Population: All participants that received study treatments, with data at the applicable post dose visit (Week 48 or Week 96). All participants received both GS010 and Sham simultaneously.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who were enrolled and received both study treatments, GS010 and Sham. Participants were randomly assigned to receive GS010 in either the right or left eye. The same participants also received the sham comparator in the eye not assigned to GS010 at the same visit.
  GS010: Either the right or left eye received one single dose of GS010 (9E10 vg/eye) via an intravitreal (IVT) injection. The volume of the injected formula was 90 µL. The injection was performed in the vitreous humor under local anesthesia.
  Sham procedure: Either the right or left eye (the eye not randomly assigned to GS010) received the sham procedure. One single sham IVT injection was performed by applying pressure to the eye at the location of a typical IVT injection procedure, using the blunt end of a syringe without a needle.
Arm/Group | All Participants
Number analyzed (Participants) | 37
Participants
  Week 48 | 37
  Week 96 | 37

5. Secondary Outcome: Change From Baseline in GCL Macular Volume at Week 48 and Week 96
Description: Ganglion cell layer (GCL) macular volume was measured as a parameter of spectral domain-optical coherence tomography (SD-OCT). SD-OCT was obtained with the Spectralis® OCT (Heidelberg Engineering).
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 36 | 36
Number analyzed (Eyes) | 36 | 36
mm^3
  Week 48 | -0.003 (0.012) | -0.038 (0.012)
  Week 96 | -0.018 (0.012) | -0.031 (0.012)

6. Secondary Outcome: Change From Baseline in RNFL Temporal Quadrant Thickness at Week 48 and Week 96
Description: Retinal nerve fiber layer (RNFL) temporal quadrant thickness was measured as a parameter of spectral domain-optical coherence tomography (SD-OCT). SD-OCT was obtained with the Spectralis® OCT (Heidelberg Engineering).
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: µm
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 36
Number analyzed (Eyes) | 37 | 36
µm
  Week 48: number analyzed (Participants) | 37 | 35
  Week 48: number analyzed (Eyes) | 37 | 35
  Week 48 | -0.562 (0.988) | -3.354 (1.017)
  Week 96: number analyzed (Participants) | 35 | 36
  Week 96: number analyzed (Eyes) | 35 | 36
  Week 96 | -1.791 (0.974) | -2.042 (0.951)

7. Secondary Outcome: Change From Baseline in Papillomacular Bundle Thickness at Week 48 and Week 96
Description: Papillomacular bundle thickness was measured as a parameter of spectral domain-optical coherence tomography (SD-OCT). SD-OCT was obtained with the Spectralis® OCT (Heidelberg Engineering).
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: µm
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 36
Number analyzed (Eyes) | 37 | 36
µm
  Week 48: number analyzed (Participants) | 37 | 35
  Week 48: number analyzed (Eyes) | 37 | 35
  Week 48 | 1.6 (1.3) | -1.0 (1.4)
  Week 96: number analyzed (Participants) | 35 | 36
  Week 96: number analyzed (Eyes) | 35 | 36
  Week 96 | 1.2 (1.3) | 0.7 (1.3)

8. Secondary Outcome: Change From Baseline in ETDRS Total Macular Volume at Week 48 and Week 96
Description: Early Treatment Diabetic Retinopathy Study (ETDRS) total macular volume was measured as a parameter of spectral domain-optical coherence tomography (SD-OCT). SD-OCT was obtained with the Spectralis® OCT (Heidelberg Engineering).
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 36 | 36
Number analyzed (Eyes) | 36 | 36
mm^3
  Week 48 | -0.104 (0.046) | -0.224 (0.046)
  Week 96 | -0.200 (0.037) | -0.265 (0.037)

9. Secondary Outcome: Change From Baseline in the Foveal Threshold Sensitivities Obtained With HVF Analyzer II at Week 48 and Week 96
Description: The assessment of standardized automated visual fields was measured using the Humphrey Visual Field (HVF) Analyzer II. Automated visual fields included the assessment of foveal threshold sensitivities. Foveal threshold sensitivity is measured in decibels (dB), which ranges from 0 dB to 50 dB. A sensitivity threshold of 0 dB indicates not being able to see the most intense perimetric stimulus, while higher dB indicates better/normal foveal vision. A positive change from baseline indicates an improvement of symptoms.
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibels (dB)
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 9 | 11
Number analyzed (Eyes) | 9 | 11
decibels (dB)
  Week 48 | 0.7 (8.9) | -0.5 (11.9)
  Week 96: number analyzed (Participants) | 8 | 9
  Week 96: number analyzed (Eyes) | 8 | 9
  Week 96 | 1.3 (8.0) | 2.4 (10.8)

10. Secondary Outcome: Visual Field Mean Deviation in Decibels of Sensitivity Obtained With HVF Analyzer II at Week 48 and Week 96
Description: The assessment of standardized automated visual fields was measured using the Humphrey Visual Field (HVF) Analyzer II. Automated visual fields included the assessment of the mean deviation (MD) in decibels (dB) of sensitivity.
Time Frame: Baseline, Week 48 and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibels (dB)
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
decibels (dB)
  Baseline MD | -25.99 (8.37) | -24.94 (9.70)
  Week 48 MD | -22.83 (9.43) | -22.94 (9.80)
  Week 96 MD | -23.22 (8.98) | -22.43 (9.39)

11. Secondary Outcome: Change From Baseline in Contrast Sensitivity at Week 48 and Week 96
Description: The assessment of contrast sensitivity was measured using the Pelli-Robson chart. The chart uses letters arranged in groups whose contrast varies from high to low. Participants read the letters, starting with the highest contrast, until they are unable to read 2 or 3 letters in a single group. Each eye is assigned a score based on the contrast of the last group in which 2 or 3 letters were correctly read, ranging from 0 to 2.2 "log of contrast sensitivity" (LogCS) units. A score of 2.0 LogCS, represents a normal sensitivity contrast, and indicates the eye was able to detect 2 of the 3 letters with a contrast of 1 percent (contrast sensitivity = 100 percent or log 2). Scores less than 2.0 signify poorer contrast sensitivity. Pelli-Robson contrast sensitivity score of less than 1.5 is consistent with visual impairment and a score of less than 1.0 represents in visual disability. A positive change from baseline indicates improvement in symptoms.
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: LogCS
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
LogCS
  Week 48 | 0.19 (0.05) | 0.09 (0.05)
  Week 96 | 0.22 (0.06) | 0.12 (0.06)

12. Secondary Outcome: Change From Baseline in Color Vision
Description: The assessment of color vision was measured using the Farnsworth-Munsell 100-Hue Color Test. Each of the 4 trays consisted of 21 caps. Participants were asked to sort the randomly arranged caps following the hue order from the first to the last fixed caps. The total error score (TES) was derived by the frequency the caps were misplaced and the severity, or distance of the misplacement.
  Errors were made whenever caps were misplaced from the correct order. Error scores were calculated according to the distance between any two caps. The error score for each individual cap was the sum of the difference between the number of that cap and the numbers of the cap adjacent to it, minus 2. TES was the total sum of the error scores of the entire set of caps.
  The best possible score was 0 and there is no defined upper limit to the total error score range. A lower score indicates improved color discrimination ability. A negative change from baseline indicates an improvement in symptoms.
Time Frame: Baseline and Week 48; Baseline and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | GS010-treated Eyes | Sham-treated Eyes
Number analyzed (Participants) | 24 | 25
Number analyzed (Eyes) | 24 | 25
score on a scale
  Week 48 | -30.0 (255.0) | -44.3 (182.2)
  Week 96: number analyzed (Participants) | 23 | 24
  Week 96: number analyzed (Eyes) | 23 | 24
  Week 96 | -10.3 (247.3) | -61.0 (188.9)

ADVERSE EVENTS:
Time Frame: From first dose to end of study (a maximum of 96 weeks)
Description: Because participants received both treatment and sham procedure simultaneously, adverse events (AEs) are reported overall for systemic and ocular AEs. Reported events include AEs associated with sham procedure.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 3/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=37)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) — This event occurred only in an eye receiving the sham procedure.
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=37)
Hypertension (Vascular disorders) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Gamma-glutamyl transferase increased (Investigations) | 8 (11)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Alcohol use (Social circumstances) | 2 (2)
Headache (Nervous system disorders) | 4 (8)
Paraesthesia (Nervous system disorders) | 2 (2)
Anterior chamber cell (Eye disorders) | 9 (11)
Autoimmune uveitis (Eye disorders) | 14 (15) — The verbatim AE term is "intermediate uveitis". 1/14 affected participants experienced this event only in sham-treated eyes.
Cataract (Eye disorders) | 4 (4) — 1/4 affected participants experienced this event only in sham-treated eyes
Conjunctival haemorrhage (Eye disorders) | 6 (7) — 3/6 affected participants experienced this event only in sham-treated eyes.
Conjunctival hyperaemia (Eye disorders) | 6 (7)
Dry eye (Eye disorders) | 2 (3) — 1/2 affected participants experienced this event only in sham-treated eyes.
Iridocyclitis (Eye disorders) | 15 (17) — 1/15 affected participants experienced this event only in sham-treated eyes.
Iritis (Eye disorders) | 2 (2)
Keratic precipitates (Eye disorders) | 13 (16)
Eye pain (Eye disorders) | 3 (4) — 1/3 affected participants experienced this event only in sham-treated eyes.
Intraocular pressure increased (Eye disorders) | 11 (13) — 1/11 affected participants experienced this event only in sham-treated eyes.
Vitritis (Eye disorders) | 6 (6)
Vitreous floaters (Eye disorders) | 2 (3)
Vitreous detachment (Eye disorders) | 2 (2)
Vitreal cells (Eye disorders) | 7 (7) — 1/7 affected participants experienced this event only in sham-treated eyes.
Visual impairment (Eye disorders) | 3 (3)
Punctate keratitis (Eye disorders) | 15 (17) — 4/15 affected participants experienced this event only in sham-treated eyes.
Depression (Psychiatric disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT02652780/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02652780/SAP_001.pdf